CLINICAL TRIAL: NCT02380443
Title: In-Situ Cancer Vaccine: Phase IIA, Open-Label Study to Assess the Safety of AlloStim® Immunotherapy Alone and in Combination With Cryoablation as Third Line Therapy for Metastatic Colorectal Cancer
Brief Title: AlloStim® Immunotherapy Dosing Alone or in Combination With Cryoablation in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirror Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITL-019-CORK-CRYVAC
Record Dates: First submitted 2015-03-02; First posted 2015-03-05 (Estimated); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2016-10

CONDITIONS: Colorectal Cancer Metastatic
Keywords: colorectal cancer; KRAS mutant; BRAF mutant; metastatic; liver metastasis; AlloStim®; cryoablation; cancer vaccine; immunotherapy; MSI-S
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dosing Schedule A (with cryoablation) (Experimental): * The priming step with ID injections of AlloStim on Days 0, 7, and 14
  * The vaccination step with cryoablation and IT (intratumoral) injection of AlloStim on Day 21
  * The activation step with IV infusion of AlloStim on Day 28
  * The booster step with two IV booster infusions of AlloStim on Days 56 and 84
  Protocol follow-up procedures continue until day 112. Efficacy evaluation will continue monthly for each subject until death or loss to follow-up
  Interventions: Biological: AlloStim; Procedure: Cryoablation
- Dosing Schedule B without cryoablation (Experimental): The priming step with ID injections of AlloStim on Days 0, 3, 7, 10 and day 14
  * IV AlloStim on Day 21
  * The booster step with two IV booster infusions of AlloStim on Days 49 and 77
  Protocol follow-up procedures continue until day 105. Efficacy evaluation will continue monthly for each subject until death or loss to follow-up Protocol follow-up procedures continue until day 105. Efficacy evaluation will continue monthly for each subject until death or loss to follow-up
  Interventions: Biological: AlloStim

INTERVENTIONS:
Biological: AlloStim — AlloStim is an activated living CD4+ Th1 memory cell derived from the blood of normal blood donors and intentionally mismatched to the recipient. AlloStim is bioengineered to express high levels of Type 1 inflammatory cytokines (such as interferon-gamma, TNF-alpha, GM-CSF) and immunomodulatory molecules such as CD40L. AlloStim has CD3/CD28-coated microbeads attached to assure activation upon infusion.
  Other Names: CryoVax
Procedure: Cryoablation — Percutaneous partial cryoablation of a single metastatic tumor lesion in the liver. The procedure is conducted under CT or ultrasound image-guidance
  Arms: Dosing Schedule A (with cryoablation)

SUMMARY:
This is a single center, open label dose frequency escalation study of CryoVax®. personalized anti-tumor vaccine protocol combining the cryoablation of a selected metastatic lesion with intra-lesional immunotherapy with AlloStim®. The in-situ (in the body) cancer vaccine step combines killing a single metastatic tumor lesion by use of cryoablation in order to cause the release of tumor-specific markers to the immune system and then injecting bioengineered allogeneic immune cells (AlloStim®) into the lesion as an adjuvant in order to modulate the immune response and educate the immune system to kill other tumor cells where ever they reside in the body.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) ranks as the third most common cancer worldwide. Metastasis is the main reason of death in CRC patients. The current drugs used to treat colorectal cancer provide important treatment options for patients, their limitations including drug resistance, poor efficacy and severe side effects. Development of new therapeutic strategies for KRAS mutant as well as BRAF mutant tumors are therefore highly needed in order to offer a new category of drug (immunotherapy). This study targets the population of mCRC patients that have progressed after two lines of chemotherapy and are not eligible for targeted therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and female subjects aged 18-80 years at screening visit
2. Pathologically confirmed diagnosis of colorectal adenocarcinoma
3. Presenting with metastatic disease:

   * Primary can be intact or previously resected
   * Metastatic lesion(s) in liver must be non-resectable
   * Extrahepatic disease acceptable
4. At least one liver lesion able to be visualized by ultrasound and determined to be safely assessable for percutaneous cryoablation
5. Previous treatment failure of two previous lines of active systemic chemotherapy:

   * Previous chemotherapy must have included an oxaliplatin-containing (e.g. FOLFOX) and an irinotecan-containing (e.g. FOLFIRI) regimen
   * with or without bevacizumab
   * administered in adjuvant setting or for treatment of metastatic disease
   * If KRAS wild type, must have at least one prior anti-EGFR therapy
   * Treatment failure can be due to disease progression or toxicity
   * Disease progression on second line therapy must be documented radiologically and must have occurred during or within 30 days following the last administration of treatment for metastatic disease
6. ECOG performance score: 0-1
7. Adequate hematological function:

   * Absolute granulocyte count ≥ 1,200/mm3
   * Platelet count ≥ 100,000/mm3
   * PT/INR ≤ 1.5 or correctable to <1.5 at time of interventional procedures
   * Hemoglobin ≥ 9 g/dL (may be corrected by transfusion)
8. Adequate Organ Function:

   * Creatinine ≤ 1.5 mg/dL
   * Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
   * Alkaline phosphatase ≤ 2.5 times ULN
   * Aspartate aminotransferase (AST) or (SGOT) ≤ 2.5 times ULN
   * Alanine aminotransferase (ALT) or (SGPT) ≤ 2.5 times ULN
9. EKG without clinically relevant abnormalities
10. Female subjects: Not pregnant or lactating
11. Patients with child bearing potential must agree to use adequate contraception
12. Study specific informed consent in the native language of the subject.

Exclusion Criteria:

1. Bowel obstruction or high risk for obstruction
2. Moderate or severe ascites requiring medical intervention
3. Clinical evidence or radiological evidence of brain metastasis or leptomeningeal involvement
4. Symptomatic asthma or COPD
5. Pulmonary lymphangitis or symptomatic pleural effusion (grade ≥ 2) that results in pulmonary dysfunction requiring active treatment or oxygen saturation <92% on room air
6. Bevacizumab (Avastin®) treatment within 6 weeks of scheduled cryoablation procedure
7. Regorafenib prior to the Study Period
8. Taking anticoagulant medication for concomitant medical condition (unless can be safely discontinued for invasive cryoablation, biopsy and intratumoral injection procedures)
9. Prior allogeneic bone marrow/stem cell or solid organ transplant
10. Chronic use (> 2 weeks) of greater than physiologic doses of a corticosteroid agent (dose equivalent to > 5 mg/day of prednisone) within 30 days of the first day of study drug treatment

    * Topical corticosteroids are permitted
11. Prior diagnosis of an active autoimmune disease (e.g., rheumatoid arthritis, multiple sclerosis, autoimmune thyroid disease, uveitis). Well controlled Type I diabetes allowed
12. Prior experimental therapy
13. History of blood transfusion reactions
14. Known allergy to bovine products
15. Progressive viral or bacterial infection

    * All infections must be resolved and the subject must remain afebrile for seven days without antibiotics prior to being placed on study
16. Cardiac disease of symptomatic nature
17. History of HIV positivity or AIDS
18. Concurrent medication known to interfere with platelet function or coagulation (e.g., aspirin, ibuprofen, clopidogrel, or warfarin) unless such medications can be discontinued for an appropriate time period based on the drug half-life and known activity (e.g., aspirin for 7 days) prior to cryoablation and biopsy procedures
19. History of severe hypersensitivity to monoclonal antibody drugs or any contraindication to any of the study drugs
20. Psychiatric or addictive disorders or other condition that, in the opinion of the investigator, would preclude study participation.
21. Subjects that lack ability to provide consent for themselves

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madappa Kundranda, MD PHD, Principal Investigator — Banner MD Anderson Cancer Center
Locations (1):
- Banner MD Anderson Medical Center, Gilbert, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epple LM, Bemis LT, Cavanaugh RP, Skope A, Mayer-Sonnenfeld T, Frank C, Olver CS, Lencioni AM, Dusto NL, Tal A, Har-Noy M, Lillehei KO, Katsanis E, Graner MW. Prolonged remission of advanced bronchoalveolar adenocarcinoma in a dog treated with autologous, tumour-derived chaperone-rich cell lysate (CRCL) vaccine. Int J Hyperthermia. 2013 Aug;29(5):390-8. doi: 10.3109/02656736.2013.800997. Epub 2013 Jun 20. PMID 23786302
- [Background] Mayer-Sonnenfeld T, Har-Noy M, Lillehei KO, Graner MW. Proteomic analyses of different human tumour-derived chaperone-rich cell lysate (CRCL) anti-cancer vaccines reveal antigen content and strong similarities amongst the vaccines along with a basis for CRCL's unique structure: CRCL vaccine proteome leads to unique structure. Int J Hyperthermia. 2013 Sep;29(6):520-7. doi: 10.3109/02656736.2013.796529. Epub 2013 Jun 4. PMID 23734882
- [Background] LaCasse CJ, Janikashvili N, Larmonier CB, Alizadeh D, Hanke N, Kartchner J, Situ E, Centuori S, Har-Noy M, Bonnotte B, Katsanis E, Larmonier N. Th-1 lymphocytes induce dendritic cell tumor killing activity by an IFN-gamma-dependent mechanism. J Immunol. 2011 Dec 15;187(12):6310-7. doi: 10.4049/jimmunol.1101812. Epub 2011 Nov 9. PMID 22075702
- [Background] Janikashvili N, LaCasse CJ, Larmonier C, Trad M, Herrell A, Bustamante S, Bonnotte B, Har-Noy M, Larmonier N, Katsanis E. Allogeneic effector/memory Th-1 cells impair FoxP3+ regulatory T lymphocytes and synergize with chaperone-rich cell lysate vaccine to treat leukemia. Blood. 2011 Feb 3;117(5):1555-64. doi: 10.1182/blood-2010-06-288621. Epub 2010 Dec 1. PMID 21123824
- [Background] Har-Noy M, Zeira M, Weiss L, Fingerut E, Or R, Slavin S. Allogeneic CD3/CD28 cross-linked Th1 memory cells provide potent adjuvant effects for active immunotherapy of leukemia/lymphoma. Leuk Res. 2009 Apr;33(4):525-38. doi: 10.1016/j.leukres.2008.08.017. Epub 2008 Oct 1. PMID 18834631
- [Background] Har-Noy M, Zeira M, Weiss L, Slavin S. Completely mismatched allogeneic CD3/CD28 cross-linked Th1 memory cells elicit anti-leukemia effects in unconditioned hosts without GVHD toxicity. Leuk Res. 2008 Dec;32(12):1903-13. doi: 10.1016/j.leukres.2008.05.007. Epub 2008 Jun 18. PMID 18565579
- [Background] Har-Noy M, Slavin S. The anti-tumor effect of allogeneic bone marrow/stem cell transplant without graft vs. host disease toxicity and without a matched donor requirement? Med Hypotheses. 2008;70(6):1186-92. doi: 10.1016/j.mehy.2007.10.008. Epub 2007 Dec 3. PMID 18054441
- [Background] Zeng Y, Stokes J, Hahn S, Hoffman E, Katsanis E. Activated MHC-mismatched T helper-1 lymphocyte infusion enhances GvL with limited GvHD. Bone Marrow Transplant. 2014 Aug;49(8):1076-83. doi: 10.1038/bmt.2014.91. Epub 2014 Apr 28. PMID 24777185

RESULTS

PARTICIPANT FLOW:
Groups:
- Dosing Schedule A (With Cryoablation): * The priming step with ID injections of AlloStim on Days 0, 7, and 14
  * The vaccination step with cryoablation and IT (intratumoral) injection of AlloStim on Day 21
  * The activation step with IV infusion of AlloStim on Day 28
  * The booster step with two IV booster infusions of AlloStim on Days 56 and 84
  Protocol follow-up procedures continue until day 112. Efficacy evaluation will continue monthly for each subject until death or loss to follow-up
  AlloStim: AlloStim is an activated living CD4+ Th1 memory cell derived from the blood of normal blood donors and intentionally mismatched to the recipient. AlloStim is bioengineered to express high levels of Type 1 inflammatory cytokines (such as interferon-gamma, TNF-alpha, GM-CSF) and immunomodulatory molecules such as CD40L. AlloStim has CD3/CD28-coated microbeads attached to assure activation upon infusion.
  Cryoablation: Percutaneous partial cryoablation of a single metastatic tumor lesion in the liver. The procedure is conducted under CT or ultrasound image-guidance
- Dosing Schedule B Without Cryoablation: The priming step with ID injections of AlloStim on Days 0, 3, 7, 10 and day 14
  * IV AlloStim on Day 21
  * The booster step with two IV booster infusions of AlloStim on Days 49 and 77
  Protocol follow-up procedures continue until day 105. Efficacy evaluation will continue monthly for each subject until death or loss to follow-up Protocol follow-up procedures continue until day 105. Efficacy evaluation will continue monthly for each subject until death or loss to follow-up
  AlloStim: AlloStim is an activated living CD4+ Th1 memory cell derived from the blood of normal blood donors and intentionally mismatched to the recipient. AlloStim is bioengineered to express high levels of Type 1 inflammatory cytokines (such as interferon-gamma, TNF-alpha, GM-CSF) and immunomodulatory molecules such as CD40L. AlloStim has CD3/CD28-coated microbeads attached to assure activation upon infusion.
Period: Overall Study
Arm/Group | Dosing Schedule A (With Cryoablation) | Dosing Schedule B Without Cryoablation
Started | 4 | 9
Completed | 3 | 9
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dosing Schedule A (With Cryoablation) | Dosing Schedule B Without Cryoablation | Total
Number analyzed (Participants) | 4 | 9 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 2 | 6 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 3 | 6 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 9 | 13
third-line MSS metastatic colorectal cancer [Count of Participants; unit: Participants] | 4 | 9 | 13

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Overall Survival
Description: Subjects are followed for survival monthly after completion of dosing
Time Frame: from time of signing informed consent for up to 18 months or until death
Measure: Median (Full Range); unit: days
Arm/Group | Dosing Schedule A (With Cryoablation) | Dosing Schedule B Without Cryoablation
Number analyzed (Participants) | 3 | 9
days | 97 [34 to 188] | 368 [184 to 440]

ADVERSE EVENTS:
Time Frame: 18 months
Description: weekly for first 90 days and monthly thereafter
Arm/Group | Dosing Schedule A (With Cryoablation) | Dosing Schedule B Without Cryoablation
All-Cause Mortality (participants affected / at risk) | 3/3 | 9/9
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/9
Other Adverse Events (participants affected / at risk) | 3/3 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dosing Schedule A (With Cryoablation) (N=3) | Dosing Schedule B Without Cryoablation (N=9)
Fatigue (Investigations) | 2 (2) | 1 (1) — Grade 3
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dosing Schedule A (With Cryoablation) (N=3) | Dosing Schedule B Without Cryoablation (N=9)
injection site reaction (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (7)
Fatigue (Investigations) | 3 (7) | 2 (3) — <grade 2
flu symptoms (Investigations) | 1 (1) | 2 (2)
pain (General disorders) | 3 (8) | 3 (3) — gastrointestinal pain
anemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) — Grade 1
edema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) — Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT02380443/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT02380443/ICF_001.pdf